CLINICAL TRIAL: NCT07106762
Title: IZABRIGHT-Bladder01: A Randomized, Open-label, Phase 2/3 Trial of Izalontamab Brengitecan Versus Platinum-based Chemotherapy for Metastatic Urothelial Cancer in Participants With Disease Progression on or After an Immunotherapy-based Treatment
Brief Title: Phase 2/3 Trial of Izalontamab Brengitecan vs Platinum-based Chemotherapy for Metastatic Urothelial Cancer With Disease Progression on or After Immunotherapy
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA244-0012; EU CTR (Other: 2025-522400-24); WHO (Other: U1111-1322-9071)
Record Dates: First submitted 2025-08-05; First posted 2025-08-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Urothelial Cancer
Keywords: Bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cisplatin; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A (Experimental)
  Interventions: Drug: Iza-bren
- Arm B (Experimental)
  Interventions: Drug: Iza-bren
- Arm C (Active Comparator)
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: Carboplatin
- Arm D (Experimental)
  Interventions: Drug: Iza-bren
- Arm E (Active Comparator)
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Iza-bren — Specified dose on specified days
  Other Names: BMS-986507; BL-B01D1; Izalontamab brengitecan
  Arms: Arm A; Arm B; Arm D
Drug: Cisplatin — Specified dose on specified days
  Arms: Arm C; Arm E
Drug: Gemcitabine — Specified dose on specified days
  Arms: Arm C; Arm E
Drug: Carboplatin — Specified dose on specified days
  Arms: Arm C; Arm E

SUMMARY:
A Phase 2/3 Trial of Izalontamab Brengitecan vs Platinum-based Chemotherapy for Metastatic Urothelial Cancer with Disease Progression on or After Immunotherapy

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed advanced urothelial carcinoma.
* Participants must be eligible to receive platinum-based chemotherapy.
* Participants must be Anti-PD-(L)1-experienced (in locally advanced or metastatic setting), either in combination with or sequential to another systemic therapy.
* Participants treated only in the peri-operative setting must have relapsed within 12 months of the last dose of the treatment.
* Participants must have ≥ 1 measurable lesion per RECIST v1.1.
* Participants must have Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.

Exclusion Criteria:

* Participants must not have platinum-based chemotherapy exposure within 12 months.
* Participants must not have received >2 prior regimens irrespective of the setting.
* Participants must not have prior ADC therapy targeting EGFR or HER3.
* Participants must not have prior therapy with topoisomerase 1 inhibitor.
* Participants must not have active, untreated brain metastases.
* Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2029-01-26 (Estimated); Study Completion 2033-11-18 (Estimated)

PRIMARY OUTCOMES:
Phase 2: Recommended Phase 3 Dose (RP3D) of BMS-986507 | Approximately 3 months
Phase 3: Progression-Free Survival (PFS) | Up to 5 years
  Assessed using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) per blinded independent central review (BICR)
Phase 3: Overall Survival (OS) | Up to 5 years

SECONDARY OUTCOMES:
Phase 2: Objective Response (OR) | Up to 5 years
  Assessed using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) by investigator
Phase 2: PFS | Up to 5 years
  Assessed using RECIST v1.1 by investigator
Phase 2: Duration of Response (DOR) | Up to 5 years
  Assessed using RECIST v1.1 by investigator
Phase 2: Time to Response (TTR) | Up to 5 years
  Assessed using RECIST v1.1 by investigator
Phase 2: OS | Up to 5 years
Phase 2: Iza-bren antibody-drug conjugate (ADC) concentration | Up to 5 years
Phase 2: Iza-bren total antibody concentration | Up to 5 years
Phase 2: Iza-bren Ed-04 payload concentration | Up to 5 years
Phase 2: Iza-bren observed concentration at end of infusion (Ceoi) | Up to 5 years
Phase 2: Iza-bren trough observed concentration (Ctrough) | Up to 5 years
Phase 3: OR | Up to 5 years
  As per RECIST v1.1 by BICR
Phase 3: DoR | Up to 5 years
  As per RECIST v1.1 by BICR
Phase 3: TTR | Up to 5 years
  As per RECIST v1.1 by BICR
Phase 3: Time until definitive deterioration in the EORTC QLQ-C30 Global Health Status/Quality of Life (GHS/QoL) scale | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (152):
- United States (32):
  - Local Institution - 0167, Gilbert, Arizona
  - Local Institution - 0162, Fullerton, California
  - Local Institution - 0252, Palo Alto, California
  - Local Institution - 0163, Sacramento, California
  - Local Institution - 0139, Sacramento, California
  - Local Institution - 0251, San Francisco, California
  - Local Institution - 0254, Santa Rosa, California
  - Local Institution - 0245, Dillon, Colorado
  - Local Institution - 0191, Edwards, Colorado
  - Local Institution - 0250, Washington D.C., District of Columbia
  - Local Institution - 0247, Miami, Florida
  - Local Institution - 0193, Lexington, Kentucky
  - Local Institution - 0232, Baltimore, Maryland
  - Local Institution - 0195, Boston, Massachusetts
  - Local Institution - 0168, Detroit, Michigan
  - Local Institution - 0248, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Local Institution - 0256, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Local Institution - 0161, Columbus, Ohio
  - Local Institution - 0257, Mayfield Heights, Ohio
  - Local Institution - 0141, Portland, Oregon
  - Local Institution - 0186, Nashville, Tennessee
  - Local Institution - 0084, Nashville, Tennessee
  - Local Institution - 0249, Abilene, Texas
  - Local Institution - 0187, Austin, Texas
  - Local Institution - 0111, Murray, Utah
  - Local Institution - 0253, St. George, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Local Institution - 0188, Norfolk, Virginia
  - Local Institution - 0200, Seattle, Washington
  - Local Institution - 0255, Seattle, Washington
- Argentina (6):
  - Local Institution - 0028, CABA, Buenos Aires
  - Local Institution - 0023, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0024, ABB, Buenos Aires F.D.
  - Local Institution - 0026, Buenos Aires, Buenos Aires F.D.
  - Local Institution - 0025, Córdoba
  - Local Institution - 0027, Mendoza
- Australia (3):
  - Macquarie University, Macquarie University, New South Wales
  - GenesisCare North Shore, St Leonards, New South Wales
  - Local Institution - 0150, Heidelberg, Victoria
- Austria (3):
  - Local Institution - 0155, Innsbruck, Tyrol
  - Medizinische Universität Wien, Vienna, Vienna
  - Local Institution - 0131, Vienna, Vienna
- Belgium (4):
  - Local Institution - 0013, Wilrijk, Antwerpen
  - AZ Maria Middelares, Ghent, Oost-Vlaanderen
  - UZ Gent, Ghent, Oost-Vlaanderen
  - Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman, Liège
- Brazil (4):
  - Local Institution - 0129, Salvador, Estado de Bahia
  - Local Institution - 0121, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0130, Rio de Janeiro
  - Local Institution - 0124, São Paulo
- Canada (4):
  - Local Institution - 0020, Edmonton, Alberta
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Local Institution - 0016, Toronto, Ontario
  - Local Institution - 0017, Montreal, Quebec
- China (24):
  - Local Institution - 0050, Beijing, Beijing Municipality
  - Local Institution - 0224, Beijing, Beijing Municipality
  - Local Institution - 0048, Fuzhou, Fujian
  - Local Institution - 0060, Fuzhou, Fujian
  - Local Institution - 0056, Xiamen, Fujian
  - Local Institution - 0051, Guangzhou, Guangdong
  - Local Institution - 0058, Guangzhou, Guangdong
  - Local Institution - 0226, Guangzhou, Guangdong
  - Local Institution - 0201, Wuhan, Hubei
  - Local Institution - 0059, Changsha, Hunan
  - Local Institution - 0044, Nanjing, Jiangsu
  - Local Institution - 0046, Nanjing, Jiangsu
  - Local Institution - 0114, Nantong, Jiangsu
  - Local Institution - 0206, Nanchang, Jiangxi
  - Local Institution - 0184, Jinan, Shandong
  - Local Institution - 0156, Qingdao, Shandong
  - Local Institution - 0205, Yantai, Shandong
  - Local Institution - 0042, Shanghai, Shanghai Municipality
  - Local Institution - 0225, Chengdu, Sichuan
  - Local Institution - 0052, Tianjin, Tianjin Municipality
  - Local Institution - 0227, Tianjin, Tianjin Municipality
  - Local Institution - 0157, Hangzhou, Zhejiang
  - Local Institution - 0053, Wenzhou, Zhejiang
  - Local Institution - 0064, Zhengzhou
- Czechia (3):
  - Local Institution - 0115, Brno, Brno-město
  - Local Institution - 0146, Hradec Králové, Hradec Králové
  - Local Institution - 0041, Prague, Praha 5
- France (12):
  - Local Institution - 0009, Nice, Alpes-Maritimes
  - Local Institution - 0040, Strasbourg, Alsace
  - CHU de Bordeaux Hop St ANDRE, Bordeaux, Aquitaine
  - Local Institution - 0006, Lyon Cedex08, Auvergne-Rhône-Alpes
  - Local Institution - 0258, Brest, Finistère
  - Local Institution - 0223, Suresnes, Hauts-de-Seine
  - Local Institution - 0002, Saint-Herblain, Loire-Atlantique
  - Local Institution - 0005, Marseille, Provence-Alpes-Côte d'Azur Region
  - Local Institution - 0003, Clermont-Ferrand, Puy-de-Dôme
  - Local Institution - 0001, Villejuif, Val-de-Marne
  - Local Institution - 0008, Paris
  - Local Institution - 0007, Paris, Île-de-France Region
- Germany (14):
  - NCT, Heidelberg, Baden-Wurttemberg
  - Local Institution - 0080, Nürtingen, Baden-Wurttemberg
  - TUM Klinikum, Munich, Bavaria
  - Klinikum Nürnberg Nord, Nuremberg, Bavaria
  - Caritas-Krankenhaus St. Josef, Regensburg, Bavaria
  - Local Institution - 0144, Hanover, Lower Saxony
  - Local Institution - 0075, Kiel, Schleswig-Holstein
  - Universitätsklinikum Jena, Jena, Thuringia
  - Local Institution - 0154, Berlin
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Krankenhaus Nordwest GmbH, Frankfurt
  - Local Institution - 0134, Hamburg
  - Marienhospital Herne, Herne
  - Universitaetsklinikum Ulm, Ulm
- Ireland (2):
  - Local Institution - 0238, Cork
  - Local Institution - 0236, Dublin
- Israel (4):
  - Local Institution - 0096, Petah Tikva, Central District
  - Local Institution - 0106, Ẕerifin, Central District
  - Local Institution - 0095, Jerusalem, Jerusalem
  - Local Institution - 0094, Haifa, Northern District
- Italy (9):
  - A.O.U.C. Policlinico di Bari, Bari, Apulia
  - Local Institution - 0107, Naples, Campania
  - Local Institution - 0099, Genoa, Liguria
  - Local Institution - 0102, Rome, Roma
  - Local Institution - 0100, Pisa, Tuscany
  - Local Institution - 0103, Padua, Veneto
  - Local Institution - 0104, Milan
  - Local Institution - 0105, Milan
  - Local Institution - 0098, Parma
- Japan (4):
  - Local Institution - 0183, Kawasaki, Kanagawa
  - Local Institution - 0171, Bunkyo-ku, Tokyo
  - Local Institution - 0169, Koto-ku, Tokyo
  - Local Institution - 0179, Toyoma, Toyama
- Netherlands (3):
  - Local Institution - 0036, Breda, North Brabant
  - Local Institution - 0033, Amsterdam, North Holland
  - Local Institution - 0031, Leeuwarden, Provincie Friesland
- Norway (3):
  - Local Institution - 0239, Lørenskog, Akershus
  - Local Institution - 0242, Tønsberg, Vestfold
  - Local Institution - 0246, Sarpsborg, Østfold fylke
- Romania (3):
  - Local Institution - 0067, Craiova, Dolj
  - Local Institution - 0066, Cluj-Napoca
  - Institutul Regional de Oncologie, Iași
- Spain (4):
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Local Institution - 0199, Valencia, Valenciana, Comunitat
  - Hospital Infanta Cristina, Badajoz
  - Hospital Universitario Virgen Del Rocio, Seville
- Sweden (3):
  - Local Institution - 0235, Solna, Stockholms Län [se-01]
  - Local Institution - 0234, Gothenburg, Västra Götalands Län [se-14]
  - Local Institution - 0241, Malmo
- Switzerland (4):
  - Cantonal Hospital St.Gallen, Sankt Gallen, Canton of St. Gallen
  - Local Institution - 0117, Bellinzona, Canton Ticino
  - Kantonsspital Graubünden, Chur
  - UniversitätsSpital Zürich, Zurich
- United Kingdom (4):
  - Local Institution - 0243, Glasgow, Glasgow City
  - St Bartholomew's Hospital, London, London, City of
  - Royal Marsden Hospital (Sutton), London, Sutton
  - Local Institution - 0230, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07106762.html